CLINICAL TRIAL: NCT01853644
Title: The Efficacy and Safety of Tivozanib in Recurrent, Platinum-Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Tivozanib in Recurrent, Platinum-Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Acronym: TIVO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Daniela Matei, Daniela Matei, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00073756
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Epithelial Ovarian Cancer; Recurrent Fallopian Tube Cancer; Recurrent Primary Peritoneal Cancer
Keywords: Cancer; Recurrent; Ovary; Fallopian Tube; Primary Peritioneal; Phase II; Platinum Resistant
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Neoplasms; Recurrence | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Tivozanib) (Experimental): Tivozanib 1.5mg orally given daily for 3 weeks with one week off to complete a 4 week cycle until disease progression or adverse effects prohibit further therapy
  Interventions: Drug: Tivozanib

INTERVENTIONS:
Drug: Tivozanib — 1.5 mg Given PO (orally)days 1-21 or every 28 day cycle
  Other Names: AV-951; Oral VEGF receptor tyrosine kinase inhibitor AV-951

SUMMARY:
This phase II trial studies how well tivozanib works in treating patients with recurrent ovarian, fallopian tube, or primary peritoneal cancer. Tivozanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical activity of tivozanib in patients with platinum-resistant, recurrent ovarian, fallopian tube or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. Determining the potential survival advantage and characterizing the safety of single agent tivozanib in patients with platinum-resistant ovarian cancer.

OUTLINE:

Patients receive tivozanib hydrochloride orally (PO) once daily (QD) on days 1-21. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must have recurrent or persistent, platinum resistant epithelial ovarian, fallopian tube or primary peritoneal carcinoma; platinum-resistant disease is defined as a recurrence within 6 months of completing adjuvant, platinum-based chemotherapy

  * Patients must have measurable disease or non-measurable (detectable) disease:

    * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be greater than or equal to 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or by clinical exam; or greater than or equal to 20 mm when measured by chest x-ray; lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI
    * Non-measurable (detectable) disease in a patient is defined in this protocol as one who does not have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria but does have a cancer antigen 125 (CA-125) greater than or equal to two times the upper normal limit within the last 60 days (confirmatory at baseline) and at least one of the following conditions:

      * Ascites and/or pleural effusion attributed to tumor
      * Hypermetabolic lesions on positron emission tomography (PET) scan
  * Patients with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST
  * Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
  * Recovery from effects of recent surgery, radiotherapy, or chemotherapy:

    * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
    * Any other prior therapy directed at the malignant tumor, including chemotherapy, biological/targeted (non-cytotoxic) agents and immunologic agents, must be discontinued at least three weeks prior to registration
    * At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy, thoracotomy, video assisted thorascopic surgery (VATS); there is no restriction on minor procedures (e.g., minor: central venous access catheter placement, ureteral stent placement or exchange, paracentesis, thoracentesis)
  * Patients must have had one prior taxane and platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organo platinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic (biologic/targeted agents, such as bevacizumab) or extended therapy administered after surgical or non-surgical assessment; there is no maximum number of prior regimens;
  * patients may not have had any prior systemic therapy (including interleukin-2, interferon-alpha, chemotherapy, bevacizumab, investigational or licensed drug that targets vascular endothelial growth factor [VEGF] or VEGF receptors/pathway or are mammalian target of rapamycin [mTOR] inhibitors) for treatment of recurrent ovarian cancer
  * Patients must have signed an approved informed consent and authorization permitting the release of personal health information
  * Patients must meet pre-entry requirements
  * A female is eligible to participate if she is of non-childbearing potential or as documentation of a negative pregnancy test prior to the start of the study treatment; sexually active pre-menopausal female subjects must agree to use adequate, highly effective contraceptive measures, while on study and for 45 days after the last dose of last study drug; effective birth control includes (a) intrauterine device (IUD) plus one barrier method; (b) oral, implantable or injectable contraceptives plus one barrier method; or (c) 2 barrier methods; effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm)

Exclusion Criteria:

* • Age < 18 years

  * Patients who have had previous treatment with tivozanib
  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count (ANC) < 1500 per mm^3
  * Platelet count < 100,000 per mm^3
  * Total bilirubin > 1.5 × upper limit of normal (ULN) (or > 2.5 x ULN for subjects with asymptomatic Gilbert's syndrome)
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN (or > 5 × ULN for subjects with liver metastasis)
  * BOTH total bilirubin > ULN AND AST/ALT > ULN
  * Alkaline phosphatase > 2.5 × ULN (or > 5 × ULN for subjects with liver or bone metastasis)
  * Creatinine > 2.0 × ULN
  * Prothrombin time (PT) such that international normalized ratio (INR) > 1.5 x ULN (unless a patient is on therapeutic warfarin) or a partial thromboplastin time (PTT) > 1.5 x ULN
  * Proteinuria > 3+ by urinalysis or urine dipstick
  * Significant cardiovascular disease, including:

    * Symptomatic left ventricular dysfunction or baseline left ventricular ejection fraction (LVEF) by multigated acquisition scan (MUGA) or echocardiogram (ECHO) of =< lower limit of institutional normal (LLN)
    * Uncontrolled hypertension: systolic blood pressure of > 140 mmHg or diastolic blood pressure of > 90 mmHg documented on 2 consecutive measurements taken at least 24 hours apart
    * Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug
    * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
    * Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
    * Coronary or peripheral artery bypass graft within 6 months of screening
    * History of class III or IV congestive heart failure, as defined by the New York Heart Association
  * Central nervous system metastases; Note: subjects with previously treated (radiotherapy or surgery) brain metastasis that have been stable without steroid treatment for at least 3 months following prior treatment may be enrolled
  * Non-healing wound, bone fracture, or skin ulcer
  * Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug
  * Serious/active infection or infection requiring parenteral antibiotics
  * Corrected QT interval (QTc) of > 480 msec using Bazett's formula
  * Radiotherapy or minor surgical procedure within 2 weeks, or major surgical procedure within 4 weeks prior to administration of first dose of study drug; inadequate recovery from prior surgical procedure
  * Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug, including but not limited to:

    * Deep vein thrombosis
    * Pulmonary embolism
    * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
    * Peripheral arterial ischemia > grade 2 (per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.0)
  * Significant bleeding disorders within 6 months prior to administration of first dose of study drug, including but not limited to:

    * Hematemesis, hematochezia, melena or other gastrointestinal bleeding >= grade 2 (per CTCAE version 4.0)
    * Hemoptysis or other pulmonary bleeding >= grade 2 (per CTCAE Version 4.0)
    * Hematuria or other genitourinary bleeding >= grade 2 (per CTCAE Version 4.0)
  * Currently active second primary malignancy, including hematologic malignancies (leukemia, lymphoma, multiple myeloma, etc.), other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast; subjects are considered to have a currently active malignancy if they have completed anti-cancer therapy and have not been disease free for > 2 years
  * Pregnant or lactating females
  * History of genetic or acquired immune suppression disease such as human immunodeficiency virus (HIV); subjects on immune suppressive therapy for organ transplant
  * Life-threatening illness or organ system dysfunction compromising safety evaluation
  * Requirement for hemodialysis or peritoneal dialysis
  * Inability to swallow capsules, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of study drugs, major resection of the stomach or small bowel, or gastric bypass procedure
  * Known hypersensitivity to drugs chemically related to tivozanib hydrochloride or sunitinib or their excipients
  * Psychiatric disorder or altered mental status precluding informed consent or protocol-related testing

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - CDH-Delnor Health System - Northwestern Medicine Cancer Center, Warrenville, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to enrollment on May 23, 2013 with the first patient being enrolled and treated on the study on June 6, 2013. The study closed to further enrollment August 10, 2018 with 31 patients registered to the study and 30 patients treated on study.
Period: Registration and Treatment Start
Arm/Group | Treatment (Tivozanib)
Started | 31
Registered | 31
Started Treatment | 30
Completed | 30
Not Completed | 1
Not completed — Did not start treatment | 1
Period: Reached First Response/Complete 2 Cycles
Arm/Group | Treatment (Tivozanib)
Started | 30
Completed | 24
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1
Not completed — Progressive Disease | 2
Period: Continued Treatment After First Response
Arm/Group | Treatment (Tivozanib)
Started | 24
Completed | 12
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Progressive Diseaes | 10
Period: Follow up for 3 Years or Until Death
Arm/Group | Treatment (Tivozanib)
Started | 30 (All patients that are treated on the study go into the follow up period)
Completed (Memo released stating that no more data to be collected after 6.10.21 for remaining patients in follow up and study is considered complete. Last follow up data collected for last patient for the study was 5.11.21.) | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the number of patients with complete response plus those with partial response as measured by RECIST 1.1 where:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Time taken to reach first best response. Range 1-4 cycles (1 cycle = 28 days)
Population: 6 patients who were determined to not be evaluable and are not included in the overall number of patients analyzed
Measure: Number; unit: participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 24
participants | 4

2. Secondary Outcome: Progression Free Survival (PFS) in Platinum-resistant Ovarian Cancer to Treatment With Single Agent Tivozanib
Description: The Kaplan-Meier method will be utilized to estimate the median and overall distribution of PFS and will be defined from the start of treatment until the first documentation of progressive disease or death, whichever occurs first..
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
months | 4.06 [1.74 to 5.78]

3. Secondary Outcome: Number of Patients Who Experienced Adverse Events in Platinum-resistant Ovarian Cancer to Treatment With Single Agent Tivozanib
Description: Adverse events will be assessed by NCI CTCAE v 4.03. Adverse event that were determined to be serious adverse events (either grade 3, 4, or 5) related to study drug were collected. Grading is as follows:In general the following severity definitions are true:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities.
  Moderate (grade 2): the event causes discomfort that affects normal daily activities.
  Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Life-threatening (grade 4): the patient was at risk of death at the time of the event. Fatal (grade 5): the event caused death.
Time Frame: During treatment and up to 30 days after completion of study treatment. Range of cycles 1-32 (1 cycle =28 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
Participants
  Hypertension | 8
  Fatigue | 3
  Hyponatremia | 2
  Colonic Fistula | 2
  Nausea | 1
  Hypomagnesemia | 1
  Anemia | 1
  Proteinuria | 1
  Hypoalbuminemia | 1
  Small intestinal perforation | 1
  Portal hypertension | 1
  Stroke | 1
  Small intestinal obstruction | 1

4. Secondary Outcome: Overall Survival (OS) in Platinum-resistant Ovarian Cancer to Treatment With Single Agent Tivozanib
Description: OS is defined from the start of treatment until date of death from any cause or date of last contact.
Time Frame: Up to approximately 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
months | 8.64 [5.39 to 12.5]

5. Post Hoc Outcome: Overall Best Response of Patients With Platinum-resistant Ovarian Cancer to Treatment With Single Agent Tivozanib
Description: Overall Best Response as measured by physical exam findings, serum CA125 levels and/or measurement of index lesions via appropriate imaging studies using RECIST criteria defined as either:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:the appearance of one or more new lesions is also considered progressions).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Time taken to reach first best response. Range 1-4 cycles (1 cycle = 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
Participants
  CR | 0
  PR | 4
  SD | 14
  PD | 6
  Not Evaluable | 6

6. Post Hoc Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the number of patients with Complete Response (CR) plus those with Partial Response (PR) plus those with Stable Disease (SD) as assessed by RECIST 1.1 where:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:the appearance of one or more new lesions is also considered progressions).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Time taken to reach first best response. Range 1-4 cycles (1 cycle = 28 days)
Population: 6 patients were determined to be not evaluable are not included in the overall number of patients analyzed
Measure: Number; unit: participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 24
participants | 18

7. Post Hoc Outcome: 3, 6, and 12 Month Progression Free Survival
Description: PFS rate will be measured by the number of patients that are progression free at 3, 6 and 12 months from treatment initiation.
Time Frame: at 3, 6 and 12 months from start of treatment
Measure: Number (95% Confidence Interval); unit: probability of patients progression free
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
probability of patients progression free
  3 months | 0.567 [0.414 to 0.775]
  6 months | 0.267 [0.147 to 0.483]
  12 months | 0.067 [0.017 to 0.254]

8. Post Hoc Outcome: Duration of Response
Description: Duration of response is defined as the time of response to the time of progression for those patients who responded. Response is generally defined as either:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: During treatment and up to 30 days after completion of study treatment. Range of cycles 1-32 (1 cycle =28 days).
Population: Only patients with a response are included
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 18
months | 5.7 [3.7 to NA] — upper limit not reached

9. Post Hoc Outcome: 3, 6 and 12 Month Overall Survival Probability
Description: OS is defined from the start of treatment until date of death from any cause or date of last contact with the probability being calculated at 3, 6 and 12 months.
Time Frame: At 3, 6 and 12 months from initiation of treatment
Measure: Number (95% Confidence Interval); unit: probability of patients alive
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 30
probability of patients alive
  3 months | 0.867 [0.753 to 0.997]
  6 months | 0.633 [0.482 to 0.832]
  12 months | 0.400 [0.258 to 0.620]

ADVERSE EVENTS:
Time Frame: AEs are collected at the beginning of every cycle (1 Cycle = 28 days) during treatment and for 30 days post last treatment. Range of cycles completed by any patient 1-32 cycles. All cause mortality data was collected during both treatment (up to 32 cycles) and follow up (up to a possible 3 years) portions of the study.
Arm/Group | Treatment (Tivozanib)
All-Cause Mortality (participants affected / at risk) | 28/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tivozanib) (N=30)
Small intestinal obstruction (Gastrointestinal disorders) | 2
Ileal obstruction (Gastrointestinal disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestinal perforation (Gastrointestinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Stroke (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tivozanib) (N=30)
Anemia (Blood and lymphatic system disorders) | 12
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 8
Anal hemorrhage (Gastrointestinal disorders) | 1
Anal stenosis (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Colonic fistula (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Oral dysesthesia (Gastrointestinal disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Fatigue (General disorders) | 15
Fever (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 8
Creatinine increased (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
INR increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 7
Weight loss (Investigations) | 9
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Obesity (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 6
Hypersomnia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 7
Proteinuria (Renal and urinary disorders) | 9
Urinary incontinence (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT01853644/Prot_SAP_000.pdf